CLINICAL TRIAL: NCT00583401
Title: Patent Foramen Ovale Closure With the AMPLATZER PFO OCCLUDER in Patients With Recurrent Cryptogenic Stroke Due to Presumed Paradoxical Embolism Through a Patent Foramen Ovale Who Have Failed Conventional Drug Therapy
Brief Title: PFO ACCESS Registry
Status: No longer available | Type: Expanded Access
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: AGA-011; G060145; NCT00557479 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2007-12-31 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Patent Foramen Ovale; Stroke
Keywords: PFO; stroke
MeSH Terms: conditions — Foramen Ovale, Patent; Stroke

INTERVENTIONS:
Device: Device closure with the AMPLATZER PFO Occluder — Device closure with the AMPLATZER PFO Occluder

SUMMARY:
Closure of Patent Foramen Ovale with the AMPLATZER® PFO OCCLUDER in patients with at least two cryptogenic strokes due to presumed paradoxical embolism through a patent foramen ovale and who have failed conventional therapy.

DETAILED DESCRIPTION:
The primary objective of the PFO Access Registry is to allow access to the AMPLATZER PFO Occluder in subjects with a PFO who have already experienced at least two cryptogenic strokes due to presumed paradoxical embolism through a patent foramen ovale and who have failed conventional drug therapy.

ELIGIBILITY:
Inclusion Criteria:

Patent foramen ovale (PFO); recurrent cryptogenic stroke; failed antiplatelet/anticoagulant therapy

Exclusion Criteria:

International normalized ration (INR) outside of 2-3; intracardiac thrombus (subjects may be enrolled after resolution of thrombus)

Sex: All
Age Groups: Child, Adult, Older Adult